CLINICAL TRIAL: NCT03401463
Title: Assesment of the Endotracheal Tube Cuff Pressure Values in ICU Pateints Before and After Training Seminar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Skladzien, MD PhD, Principal Investigator, Jagiellonian University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1072.6120.194.2017
Record Dates: First submitted 2018-01-03; First posted 2018-01-17 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Respiratory Tract Diseases; Respiratory Tract Infections; Pneumonia, Ventilator-Associated; Ventilator-Induced Lung Injury
Keywords: endotracheal tube cuff pressure; Ventilator-Induced Lung Injury; traning
MeSH Terms: conditions — Respiratory Tract Diseases; Respiratory Tract Infections; Pneumonia, Ventilator-Associated; Ventilator-Induced Lung Injury

STUDY DESIGN:
Intervention Model Description: The study will include patients staying in the intensive care unit, requiring ventilation of the artificial airways in the form of endotracheal or tracheostomy tube. Patients will be over 18 years of age.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- once a day (Active Comparator): Cuff pressure checks once a day.
  Interventions: Other: traning seminar
- three times a day (Active Comparator): Cuff pressure checks three times a day
  Interventions: Other: traning seminar

INTERVENTIONS:
Other: traning seminar — There will be provided 30 min training seminar on the function of endotracheal cuff and cuff pressure.

SUMMARY:
There is no accepted standard for the frequency of monitoring endotracheal tube cuff pressures (ETCP). the investigators plan on comparing two strategies for monitoring ETCP in mechanically ventilated patients.

Nowadays ETCP is evaluated once every 24 hours. Next, the investigator want to conduct training for medical and nursing staff. After the training, ETCP will be measured every 8 hours.

The aim of the study is to prove that more frequent pressure control (3 times a day) reduces the occurrence of abnormal ETCP.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated patients intubated in a medical intensive care unit

Exclusion Criteria:

* Patient requiring prone positioning, tracheo-esophageal fistula, lung transplant and neutropenic patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
monitoring of cuff pressures | 1 year
  The effectiveness of pressure monitoring in various time intervals

SECONDARY OUTCOMES:
preventing complications of incorrect pressure in tracheal cuff | 5 years
  preventing of an VAP or airway damage

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Undecided
We are undecided on this point.